CLINICAL TRIAL: NCT05110274
Title: Validating a Novel Approach to Assess Metabolic Flexibility in a Respiratory Chamber
Acronym: METFLEX II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, David McDougal, Assistant Professor - Research, Pennington Biomedical Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PBRC 2021-031
Record Dates: First submitted 2021-10-04; First posted 2021-11-05 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sequential measurements of metabolic flexibility (Experimental): Study participants will undergo three assessments of metabolic flexibility. Two measurements of metabolic flexibility will be conducted during two separate overnight stay in a metabolic chamber approximately 5-7 days apart. The third measurement of metabolic flexibility will be assessed during a hyperinsulinemic-euglycemic clamp procedure conducted 7-28 days following the completion of the second overnight stay in the metabolic chamber.
  Interventions: Procedure: Overnight Metabolic Flexibility; Procedure: Clamp Metabolic Flexibility

INTERVENTIONS:
Procedure: Overnight Metabolic Flexibility — Participants will spend 13 hours (overnight) in a metabolic chamber where they will be fed a single high-fat supper meal. Energy expenditure, respiratory exchange ratio (RER), and 12-h oxidation of CHO, fat, and protein will be calculated and used to determine metabolic flexibility, i.e. change in RER from baseline.
Procedure: Clamp Metabolic Flexibility — Metabolic flexibility with be assessed during a 2-step hyperinsulinemic-euglycemic clamp procedure. The clamp will be performed for four hours, two hours at an insulin dose of 10 mU/m^2/min and two hours at an insulin dose of 80 mU/m^2/min. Resting metabolic rate will be determined via hood indirect calorimetry at baseline, before insulin onset, and during the final 30 min of each step of the clamp. Metabolic flexibility will be determined by comparing the resting metabolic rate during baseline and during the final 30 min of each step of the clamp.

SUMMARY:
This study is designed to test the reliability of a novel procedure for measuring metabolic flexibility, i.e., the ability to quickly adapt macronutrient oxidation to macronutrient availability, in a respiratory chamber. The investigators will compare paired measurements of metabolic flexibility determined 5-7 days apart in a metabolic chamber to assess reliability. The investigators will also compare their novel method of measuring metabolic flexibility in a respiratory chamber with a more convention method, metabolic flexibility during a hyperinsulinemic clamp.

DETAILED DESCRIPTION:
Metabolic flexibility (METFLEX) is the ability to adapt fuel oxidation to fuel availability and energy demands. Impaired METFLEX is associated with weight gain, ectopic lipid deposition, insulin resistance, and the potential development of type 2 diabetes. Even if impaired METFLEX shows promise as an early predictor of future metabolic dysfunction, longitudinal studies have been lacking because of the absence of simple methods for assessing METFLEX. This project will further validate (reproducibility and comparison with hyperinsulinemic-euglycemic clamps) a novel approach for measuring METFLEX recently developed by the PI.

METFLEX is commonly measured during a hyperinsulinemic-euglycemic clamp. Yet, this technique is questioned because it relies on a non-physiological stimulus (intravenous glucose and insulin) and inherently suppresses fat oxidation via non physiological hyperinsulinemic conditions. In contrast, impaired fat oxidation in response to a high-fat meal is a more physiological indicator of metabolic inflexibility. The investigators have recently developed a method for measuring METFLEX by assessing the dynamics in respiratory exchange ratio (RER) in response to a high-fat standardized dinner in a whole-body room indirect calorimeter. Securing extramural funding for the aforementioned longitudinal studies employing this novel methodology is presently limited due to a lack of the following preliminary data: 1) quantification of the intra-subject variability of this novel METFLEX measure to perform power calculations (sample size) in large-scale prospective clinical trials, and 2) comparison of our method to a more accepted measurement of METFLEX. The overarching goal of this method development project is to generate reproducibility and validity data of The investigators' new assessment of METFLEX in a whole-body room indirect calorimeter against the METFLEX measured by a hyperinsulinemic-euglycemic clamp.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5 kg/m^2 and 35 kg/m^2 (±0.5 kg/m^2 will be accepted)
* Willing to consume pre-prepared meals
* Non pregnant
* Bilateral oophorectomy or use of the following contraceptive methods (females only):

  1. monophasic oral contraceptives
  2. progesterone-only oral contraceptives
  3. injectable or implantable progesterone-only contraceptives

Exclusion Criteria:

* Unstable weight in the last 3 months [gain or loss >7 lb (or 3.2 kg)]
* Currently working shift work
* Smoking or use of tobacco products within the last 3 months
* History of clinically diagnosed diabetes or a fasting blood glucose >126 mg/dL
* Average screening blood pressure >140/90 mmHg
* Previous bariatric surgery (or other surgeries) for obesity or weight loss
* Use of medications affecting metabolism or sleep**
* History of cardiovascular disease, neurological disease, or other chronic diseases that affect sleep or metabolism
* Pregnant, planning to become pregnant, or breastfeeding
* Adherence to special restrained diets (e.g., low-carbohydrate, low-fat, or vegetarian/vegan diets) over the last 3 months.

  * Sporadic use of these medications is acceptable (however, enrollment will be evaluated on a case-by-case basis). If taking sporadically, participants should not be taking the medication for 1-month prior to the first visit.

NOTE: Participants may also be excluded if deemed medically necessary by study Medical Investigator.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
peak decrease in overnight respiratory exchange ratio | 12 hours
  mean of peak decrease in respiratory exchange ratio (baseline values -nadir values) following the test meal during an overnight stay in a respiratory chamber.
  Peak values are defined as the lowest respiratory exchange ratio value measured during the sleep period, 11pm-5am
  Baseline values are measured 1h prior to meal (5:00-5:45pm)
  An increase in this value indicates increased metabolic flexibility.
change in respiratory exchange ratio during high-dose insulin infusion | 4.5 hours
  mean of peak increase in respiratory exchange ratio during a 80 mU/m^2/min insulin infusion (insulin stimulated - baseline values) that is conducted during an hyperinsulinemic-euglycemic clamp procedure..
  Insulin-stimulated values are defined as the mean respiratory exchange ratio value measured during the final 30 min of a 2 hour 80 mU/m^2/min insulin infusion.
  Baseline values are measured 30 min prior to the start of the hyperinsulinemic-euglycemic clamp procedure.
  An increase in this value indicates increased metabolic flexibility.

SECONDARY OUTCOMES:
slope of respiratory exchange ratio | 12 hours
  This value indicates the speed and magnitude of the participants change in respiratory exchange ratio between the peak and nadir values measured overnight in the respiratory chamber.
  A more negative value in this measurement indicates either a short time interval between the highest and lowest respiratory exchange ratio values measured and/or a large difference between the highest and lowest values of respiratory exchange ratio values measured.
respiratory exchange ratio/food quotient (RER:FQ ratio) | 12 hours
  The ratio of the 12-h respiratory exchange ratio to the food quotient of the meal.
  This measurement assesses the degree to which a participant's actual respiratory exchange ratio matches the theoretical respiratory exchange ratio that would be obtained if all the macronutrients in the test meal were oxidized during an overnight stay in a respiratory chamber.
  A value of 1 indicates perfect agreement between measured and theoretical values. A value greater than 1 indicates a lack of fat oxidation, while a value less than 1 indicates a lack of carbohydrate oxidation.
  Individuals with high metabolic flexibility should achieve values closer to 1 than individuals with low metabolic flexibility.
change in respiratory exchange ratio during low-dose insulin infusion | 4.5 hours
  mean of peak increase in respiratory exchange ratio during a 10 mU/m^2/min insulin infusion (insulin stimulated - baseline values) that is conducted during an hyperinsulinemic-euglycemic clamp procedure..
  Insulin-stimulated values are defined as the mean respiratory exchange ratio value measured during the final 30 min of a 2 hour 10 mU/m^2/min insulin infusion.
  Baseline values are measured 30 min prior to the start of the hyperinsulinemic-euglycemic clamp procedure.
  An increase in this value indicates increased metabolic flexibility.
Time to nadir respiratory exchange ratio | 12 hours
  Average time from meal to nadir respiratory exchange ratio value
  This measurement indicates how long on average it took form the onset of the meal, 6pm, for the participants to achieve their lowest/nadir respiratory exchange ratio value during an overnight stay in a respiratory chamber..
Time to food quotient | 12 hours
  Average time from meal to a participant's respiratory exchange ratio reaching the food quotient of the test meal
  This measurement indicates how long on average it takes form the onset of the meal, 6pm, for the participants to register a respiratory exchange ratio equal to the food quotient of the test meal during an overnight stay in a respiratory chamber.
  A reduction in this value indicates increased metabolic flexibility.

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States